CLINICAL TRIAL: NCT05530928
Title: The Importance of Including Reproductive Life Plan Counseling During Contraceptive Counseling: a Randomized Controlled Trial
Brief Title: The Importance of Including Reproductive Life Plan Counseling During Contraceptive Counseling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: Tfem/2022'/23
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Family Planning Services
Keywords: Preconception health; Reproductive life plan; Family planning

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will receive the standard care (standard family planning counseling)
- Intervention Group (Other): This group will receive the standard family planning counseling + reproductive life plan counseling.
  Interventions: Other: Reproductive life plan counseling

INTERVENTIONS:
Other: Reproductive life plan counseling — The intervention group will receive in addition to the standard contraceptive counseling, a reproductive life plan counseling: midwives will discuss the different options with the woman depending if she wants or not more children, and she will give her general information about preconception health.
  Arms: Intervention Group

SUMMARY:
The reproductive life plan is a protocol intended to promote preconception planning, improve reproductive health and increase health knowledge. The aim of the study is to evaluate the importance of including the reproductive life plan counseling during contraceptive counseling.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the outcomes of the reproductive life plan counseling on knowledge about fertility and awareness of preconception health.

2 groups of women visiting a primary health care center for contraceptive counseling are formed: a control group that will receive the standard care (standard family planning counseling) and the intervention group that will receive the standard family planning counseling in addition to the reproductive life plan counseling.

The included women are aged between 20 and 40 years. They are informed about the study when they call the center to make their appointment. When they attend the center, they receive a written and oral information and they are also informed that participation is voluntary and that they can interrupt their participation at any time without explanation. The women who agree to participate will sign an informed consent.

The midwives will be trained to reproductive life plan counseling before the commencement of the study. They have access to a template with discussion points to choose from, depending on the woman's answer to the first question (Do you want children/more children in the future?). If the answer is "no" the counseling will focus on contraceptive methods and sexual health (avoiding sexually transmitted diseases). If the answer is "yes" the discussion will focus on preconception and reproductive health (avoiding alcohol and tobacco, taking folic acid at least one month before conception, avoiding under and overweight,...).

Randomization: sealed envelopes are prepared with notes for CG (control group) or IG (intervention group). Before starting the counseling, the midwife opens the envelope containing instructions for either CG or IG.

A questionnaire is filled by the women before starting the counseling session and another one 2 months after the intervention. The questionnaire contains questions about demographics, knowledge about fertility, preconception health and the use of contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 40 years old visiting the health center

Exclusion Criteria:

* Women that refuse to participate in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 164 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge about fertility | 2 months
  Unit of measure: The percentage of women who answer correctly the questions about fertility.
  Measurement tool: Questionnaire using the following questions (probability of a 25-year-old woman becoming pregnant if she had unprotected intercourse, fecundity time of an ovum, the age of decline of woman's fertility, the chance of giving birth after in-vitro fertilization).
  This outcome is compared between the intervention group and the control group.
Awareness of preconception health | 2 months
  Unit of measure: The percentage of women who answer correctly the questions about preconception health.
  Measurement tool: Questionnaire using the following questions (the importance for a woman to stop using tobacco, to refrain from alcohol, to be of normal weight, and to start with folic acid before a pregnancy).
  This outcome is compared between the intervention group and the control group.

SECONDARY OUTCOMES:
The use of contraception | 2 months
  Unit of measure: The percentage of women who used contraceptive methods during their latest sexual intercourse.
  Measurement tool: Questionnaire through questions about the usage of different contraception methods.

CONTACTS AND LOCATIONS:
Locations (2):
- Lebanon (2):
  - Contraceptive service center, Bekaa
  - Contraceptive service center, Tyre

IPD SHARING:
Plan to Share IPD: No